CLINICAL TRIAL: NCT07367425
Title: Risks of Ramadan Fasting in Patients With Primary Adrenal Insufficiency Treated With Prednisolone.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital La Rabta (Other)
Responsible Party: Principal Investigator, Melika Chihaoui, Professor of Endocrinology, Faculty of Medicine of Tunis, University Tunis El Manar. Head of the Department of Endocrinology, University hospital La rabta, Tunis, Tunisia., Hopital La Rabta
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: HLaRabta26
Record Dates: First submitted 2026-01-16; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Primary Adrenal Insufficiency; Ramadan Fasting; Prednisolone; Continuous Glucose Monitoring; Hypoglycemia Non-Diabetic; Dehydration
Keywords: primary adrenal insufficiency; Ramadan fasting; continuous glucose monitoring; hypoglycemia; dehydration; glucocorticoid replacement therapy; prednisolone; hypotension
MeSH Terms: conditions — Addison Disease; Dehydration; Hypoglycemia; Hypotension

STUDY DESIGN:
Intervention Model Description: The study of patients with PAI treated with prednisolone 5mg/day for 14 days before fasting, then during 14 days of Ramadan fasting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Outside Ramadan fasting (No Intervention): Patients with PAI treated with prednisolone 5mg/day, outside Ramadan fasting
- Ramadan fasting (Experimental): Patients with PAI treated with prednisolone 5mg/day during Ramadan fasting.
  Interventions: Other: Ramadan fasting

INTERVENTIONS:
Other: Ramadan fasting — Ramadan fasting is a religious dry intermittent fasting
  Other Names: dry intermittent fasting
  Arms: Ramadan fasting

SUMMARY:
In primary adrenal insufficiency (PAI), there is a risk of hypoglycemia and dehydration. These risks seem to be increased during intermittent fasting. A previous study in patients with PAI treated with hydrocortisone at a dose of 20 mg/day showed that the prevalence of hypoglycemia was as high outside (63%) as during Ramadan fasting (71%), and that there was no risk of dehydration. We propose to evaluate the risk of complications during and outside of Ramadan fasting through a prospective study with subjects taken as their own controls, in 35 patients with PAI treated with prednisolone at a dose of 5 mg/day. Patients will undergo an interview, physical examination, blood sampling, and continuous glucose monitoring (CGM) during two weeks of fasting and two weeks of non-fasting.

DETAILED DESCRIPTION:
The risk of hypoglycemia in adrenal insufficiency is known but poorly studied. It is due to cortisol deficiency. Only a few publications have addressed this topic. The risk of hypoglycemia is thought to be increased during acute decompensation, following treatment discontinuation, and during fasting or delayed eating. Thus, this risk is thought to be increased during intermittent fasting, such as the Ramadan fast. A previous study conducted in the endocrinology department of La Rabta Hospital, involving 30 subjects with corticotropic insufficiency who underwent 24-hour continuous glucose monitoring (CGM), identified three cases of hypoglycemia during intermittent fasting and no hypoglycemia outside of fasting periods. A more recent study showed that the prevalence of hypoglycemia, assessed by a seven day-CGM, was 63% outside of fasting and 71% during Ramadan fasting in subjects with PAI substituted with hydrocortisone at the usual dose of 20mg/day.

The most commonly used glucocorticoid replacement therapy is based on hydrocortisone or cortisone. Prednisolone is also indicated, particularly in cases difficult to control with hydrocortisone. The usual dose is 5 mg/day. It has been suggested to replace hydrocortisone with prednisolone to reduce the risk of complications during Ramadan fasting. However, this has never been demonstrated. A previous study showed that the prevalence of complications, quality of life, and point-in-time capillary blood glucose measurements were not different with hydrocortisone or prednisolone.

On the other hand, the risk of dehydration and hypotension seems to be low in patients treated with hydrocortisone.

General objective:

To evaluate the risks of intermittent fasting in subjects with PAI treated with prednisolone 5 mg/day.

Specific objectives:

* To evaluate the frequency of hypoglycemia in subjects with PAI treated with prednisolone 5 mg/day during and outside of Ramadan fasting.
* To evaluate the frequency of dehydration in subjects with PAI treated with prednisolone 5 mg/day during and outside of Ramadan fasting.
* To study the factors associated with hypoglycemia and dehydration.

Study type: prospective, interventional, with the subject serving as their own control.

Visit 1: 4 weeks before Ramadan

* Verification of inclusion and exclusion criteria.
* Explanation of the study objectives and procedures.
* Obtaining informed consent from the patient.
* Switching from hydrocortisone to prednisolone 5 mg/day. Fludrocortisone will be continued, and the dose will be adjusted if necessary.

Visit 2: 14 days before Ramadan, patients treated with prednisolone for 14 days.

This visit will include an interview, a physical examination, placement of a CGM system, and a fasting blood sample.

Interview:

* Demographic data: age, sex
* Data related to PAI: duration, etiology, replacement therapy. History of fasting and its duration (number of days fasted, occurrence of complications).
* Quality of life questionnaire (AddiQoL) and sleep quality questionnaire (PSQI). Physical examination: weight, height, waist circumference, blood pressure (lying and standing), heart rate, presence of hyperpigmentation, signs of dehydration.

The CGM device, consisting of a subcutaneous sensor (2.5 mm flexible catheter) and a transmitter (single-use), will be inserted. This device measures and records interstitial glucose every three minutes for 14 days.

The CGM application will be downloaded to the patient's or a parent's smartphone for data collection and transmission.

* Issuance of monitoring sheets. During the 14 days of CGM, patients will be required to complete a monitoring sheet including medication intake, wake-up and bedtimes, physical activity, and any adverse events (fatigue, signs of hypoglycemia, signs of hypotension, or other symptoms). Patients will be contacted by one of the investigators by telephone to ensure adherence to the protocol and to monitor for any potential complications.
* Laboratory tests: urea, electrolytes.

Visit 3: During Ramadan (the first 14 days). This visit will include an interview, a physical examination, placement of the CGM device, and a fasting blood sample, following the same procedure as Visit 2.

* The patient will receive dietary and lifestyle advice regarding fasting.
* Monitoring forms will be provided. During this study period, patients will also be required to complete the same monitoring form. Patients will also be contacted by one of the investigators by telephone to verify adherence to the protocol and to monitor for any potential complications.

The criteria for breaking the fast are:

Occurrence of discomfort during fasting, hypoglycemia on MCG, elevated urea, or hyperkalemia.

Visit 4: After Ramadan, patients should submit their monitoring records.

Diagnostic criteria:

* First-degree hypoglycemia is defined as an interstitial glucose level measured during continuous glucose monitoring (CGM) < 0.70 g/L for more than 15 minutes, and second-degree hypoglycemia as an interstitial glucose level < 0.55 g/L for more than 15 minutes.
* Dehydration is defined by the onset of arterial hypotension (BP < 90/60 mmHg or orthostatic hypotension) or an elevation of plasma urea.

Statistical analysis:

The frequencies of hypoglycemia and dehydration will be calculated and compared between the fasting and non-fasting periods. Mean blood glucose levels per period (suhoor-5 a.m.; 5 a.m.-10 a.m.; more than 10 a.m. after suhoor) will also be calculated and compared between the fasting and non-fasting periods. Univariate and potentially multivariate analyses will be conducted to determine the factors associated with hypoglycemia and dehydration.

ELIGIBILITY:
Inclusion Criteria:

* subjects with primary adrenal insufficiency known for at least one year, treated with a glucocorticoid and a mineralocorticoid, who wish to fast during Ramadan 2026.

Exclusion Criteria:

* presence of diabetes, renal, hepatic, cardiac, or respiratory insufficiency; use of hypoglycemic agents (sulfonylureas), diuretics, use of any glucocorticoid other than the prescribed replacement therapy; poor disease control (asthenia, malaise, hyperpigmentation, discontinuation of treatment, etc.); pregnancy; breastfeeding; menstruation.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2026-01-22 (Estimated); Primary Completion 2026-03-22 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Hypoglycemia | during 14 days before Ramdan fasting and 14 days of Ramdan fasting
  Diagnosed using continuous glucose monitoring
Dehydration | During the 14 days before Ramadan fasting and during the 14 days of Ramadan fasting.
  Hypotension and increased serum urea

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital La Rabta, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided
IPD can be shared with other researchers on a reasonable request.

REFERENCES:
- [Background] Chihaoui M, Yazidi M, Oueslati I, Khessairi N, Chaker F. Intermittent fasting in adrenal insufficiency patients: a review and guidelines for practice. Endocrine. 2021 Oct;74(1):11-19. doi: 10.1007/s12020-021-02804-z. Epub 2021 Jul 2. PMID 34213700
- [Background] Hussain S, Hussain S, Mohammed R, Meeran K, Ghouri N. Fasting with adrenal insufficiency: Practical guidance for healthcare professionals managing patients on steroids during Ramadan. Clin Endocrinol (Oxf). 2020 Aug;93(2):87-96. doi: 10.1111/cen.14250. Epub 2020 Jun 15. PMID 32419166
- [Background] Chihaoui M, Mimita W, Oueslati I, Rejeb O, Ben Amor Z, Grira W, Yazidi M, Chaker F. Prednisolone or hydrocortisone replacement in patients with corticotrope deficiency fasting during Ramadan result in similar risks of complications and quality of life: a randomized double-blind controlled trial. Endocrine. 2020 Jan;67(1):155-160. doi: 10.1007/s12020-019-02082-w. Epub 2019 Sep 24. PMID 31552584
- [Background] Chihaoui M, Sta J, Kamoun E, Belhadjsliman C, Khessairi N, Oueslati I, Yazidi M, Chaker F, Feki M. Hypoglycaemia and other risks of ramadan fasting in patients with primary adrenal insufficiency: A prospective controlled trial using 24-hour glucose monitoring. J Endocrinol Invest. 2025 Oct 18. doi: 10.1007/s40618-025-02728-9. Online ahead of print. PMID 41108503
- [Background] Chihaoui M, Grira W, Bettaieb J, Yazidi M, Chaker F, Rejeb O, Oueslati I, Feki M, Kaabachi N, Slimane H. The risk for hypoglycemia during Ramadan fasting in patients with adrenal insufficiency. Nutrition. 2018 Jan;45:99-103. doi: 10.1016/j.nut.2017.07.014. Epub 2017 Aug 3. PMID 29129244